CLINICAL TRIAL: NCT06520033
Title: Robotics as a Useful Tool to Improve the Hydration of the Elderly
Acronym: Hidroponent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Collaborators: Agency for Management of University and Research Grants (Catalonia, Spain) (Unknown); Hospital Universitari Santa Maria (Lleida, Spain) (Unknown)
Responsible Party: Principal Investigator, Teresa Botigué Satorra, Principal Investigator, Universitat de Lleida
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N23059; 2023 CLIMA 00047 (Other Grant/Funding Number: Agency for Management of University and Research Grants)
Record Dates: First submitted 2024-06-26; First posted 2024-07-25 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Dehydration; Daily Fluid Intake; Urinary Infections
Keywords: dehydration; aged; nursing homes; robotics; fluid intake
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive a hydration plan executed by a humanoid robot.
  Healthcare personnel will receive reminders from the robot to record fluid intake through it.
  Interventions: Device: humanoid robot
- Control group with (Active Comparator): The control group will receive the center's usual hydration plan. The health personnel will make the fluid intake record in paper format and at the end of the shift, as usual.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: humanoid robot — The humanoid robot will execute an educational hydration plan that will be integrated into the usual dynamics of the residence. In order to increase the fluid intake of the residents, stimulation activities will be proposed that will be carried out by the robot such as reminders, interactive activities and positive reinforcement. It will also allow the daily recording fluid intake of each residents.
  This intervention will last two months.
  Arms: Intervention group
Other: Usual care — The center's usual hydration plan
  Arms: Control group with

SUMMARY:
The aim of this clinical trial is to evaluate the effectiveness of a hydration educational program executed through a robot in comparison with the usual hydration program in terms of fluid intake and general health status of the residents. The main question to be answered is whether the use of robotics through a humanoid robot increases the hydration of institutionalized older people.

Participants:

* The intervention group will receive a hydration plan executed by the robot and the control group will receive the center's usual hydration plan.
* Healthcare personnel will receive reminders from the robot to record fluid intake through it. In the control group, health personnel will perform the fluid intake record in paper format and at the end of the shift, as usual.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 65 years.

No exclusion criteria have been established.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 57 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Daily fluid intake | From enrollment to the end of intervention at 8 weeks
  Amount in milliliters (ml)
Urine color | 8 weeks
  Urine color chart (Armstrong, 2000). Values = 1 - 8. Dehydration: scores >= 4
Serum osmolarity | 8 weeks
  Serum osmolarity: [1,86*(Na+K)+1,15*Glucose+urea+14)]. Dehydration > 300mOsm/kg
Blood Urea Nitrogen | 8 weeks
  BUN = Urea/2.1428. Dehydration > 20mg/dl
Number of urinary infections | 8 weeks
  Obtained through a urine sample and evaluated with the Combur-Test.

SECONDARY OUTCOMES:
Dry Skin | 8 weeks
  Skin turgor: if skin remains elevated after being pulled up and released
Cognitive status | 8 weeks
  The Mini Cognitive Examination (MEC) (Values = 0 - 30). Cognitive impairment: scores <= 23
Cognitive status | 8 weeks
  Global Deterioration Scale (GDS). Values = 1 - 7. Dementia: scores >= 3
Risk of falls | 8 weeks
  Downton scale. Values = 0 - 11. Risk of falls: scores > 2
Illnesses | 8 weeks
  Diseases that the participant currently presents
Pharmacological treatment | 8 weeks
  Number of medicines taken by the participant per day and type of medicine.
Efficacy and safety of swallowing | 8 weeks
  Volume-Viscosity swallow test (V-VST): identify clinical signs of impaired efficacy (labial seal, oral and pharyngeal residue, and piecemeal deglutition) and impaired safety of swallow (voice changes, cough and decrease in oxygen saturation ≥3%). It starts with nectar viscosity and increasing bolus volume, then liquid and finally pudding viscosity
Nutritional status | 8 weeks
  Assessed through the Mini Nutritional Assessment (MNA). Values = 0 - 30. Malnutrition: scores < 17
Risk of pressure ulcers | 8 weeks
  Braden Scale. Values = 6 - 23. Risk of pressure ulcers: scores < 19
Functional status | 8 weeks
  Barthel index. Values = 0 - 100. Functional impairment: scores < 90
Hospital admissions | 8 weeks
  Number of hospital admissions

OTHER OUTCOMES:
Education level | Baseline
  Choose between: no studies, primary studies, secondary studies and university studies.
Birthdate | Baseline
  Date of birth in yyyy/mm/dd format
Marital status | Baseline
  The answer options are: single, married, in partnership (but not married), separated or divorced (currently without a partner), widow (If the answer is "yes"must be specified if less than one year or not).
Date of institutionalization | Baseline
  Date in yyyy/mm/dd format when the resident began to be institutionalized in the center.
Sex | Baseline
  Female or male sex

CONTACTS AND LOCATIONS:
Locations (1):
- Residència i Centre de Dia per a Gent Gran Balàfia II, Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Botigue T, Miranda J, Escobar-Bravo MA, Lavedan A, Roca J, Masot O. [Analysis of dehydration in older people in a nursing home in Spain: prevalence and associated factors]. Nutr Hosp. 2021 Apr 19;38(2):252-259. doi: 10.20960/nh.03260. Spanish. PMID 33593070
- [Background] Masot O, Miranda J, Santamaria AL, Paraiso Pueyo E, Pascual A, Botigue T. Fluid Intake Recommendation Considering the Physiological Adaptations of Adults Over 65 Years: A Critical Review. Nutrients. 2020 Nov 4;12(11):3383. doi: 10.3390/nu12113383. PMID 33158071
- [Background] Botigue T, Masot O, Miranda J, Nuin C, Viladrosa M, Lavedan A, Zwakhalen S. Prevalence and Risk Factors Associated With Low Fluid Intake in Institutionalized Older Residents. J Am Med Dir Assoc. 2019 Mar;20(3):317-322. doi: 10.1016/j.jamda.2018.08.011. Epub 2018 Oct 15. PMID 30337227
- [Background] Masot O, Iglesias Millan A, Nuin C, Miranda J, Lavedan A, Botigue T. [How to improve hydration and fluid intake in institutionalized older people? A scientific literature review]. Nutr Hosp. 2018 Dec 3;35(6):1441-1449. doi: 10.20960/nh.1885. Spanish. PMID 30525860
- [Background] Masot O, Lavedan A, Nuin C, Escobar-Bravo MA, Miranda J, Botigue T. Risk factors associated with dehydration in older people living in nursing homes: Scoping review. Int J Nurs Stud. 2018 Jun;82:90-98. doi: 10.1016/j.ijnurstu.2018.03.020. Epub 2018 Mar 27. PMID 29626702